CLINICAL TRIAL: NCT02245009
Title: Safety of External Electrocardioversion in Device Patients - the SEED Registry
Brief Title: Safety of External Electrocardioversion in Device Patients
Acronym: SEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: UKK-SEED-2014
Record Dates: First submitted 2014-09-05; First posted 2014-09-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Atrial Arrhythmia
MeSH Terms: interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Pacemaker patients: Patients with pacemaker, presenting for cardioversion.
  Interventions: Procedure: Cardioversion
- ICD patients: Patients with ICD, presenting for cardioversion.
  Interventions: Procedure: Cardioversion
- CRT patients: Patients with CRT device, presenting for cardioversion.
  Interventions: Procedure: Cardioversion

INTERVENTIONS:
Procedure: Cardioversion

SUMMARY:
Arrhythmias of the atria of the heart are a common comorbidity in patients with cardiac rhythm management devices, such as pacemakers and implantable cardioverter/defibrillators (ICD). External electrical cardioversion is an established method to achieve rhythm control (restore normal sinus rhythm) in patients with atrial arrhythmia. Little data on safety and efficacy of external electrical cardioversion in patients with cardiac rhythm management devices exists. Thus, available data on the safety of external electrical cardioversion in cardiac rhythm management patients lacks statistical power to accurately reflect the true hazard of external electrical cardioversion in patients with cardiac rhythm management devices.

The aim is to systematically include and follow all patients with cardiac rhythm management devices presenting for external electrical cardioversion, to analyse the effects of external electrical cardioversion on leads and devices.

DETAILED DESCRIPTION:
Introduction Atrial arrhythmias are a common comorbidity in patients with cardiac rhythm management (CRM) devices, such as pacemakers and ICD. External electrical cardioversion is an established method to achieve rhythm control in patients with atrial arrhythmia. A paucity of data on safety and efficacy of external electrical cardioversion in patients with cardiac rhythm management devices exists. Most publications are of older date and predominantly case reports or case collections. Few prospective studies with a population of cardiac rhythm management patients after external electrical cardioversion have been published in recent years.

Thus, available data on the safety of external electrical cardioversion in cardiac rhythm management patients lacks statistical power to accurately reflect the true hazard of external electrical cardioversion in patients with cardiac rhythm management devices.

Rationale Electrocardioversion in Propofol sedation for atrial or ventricular tachyarrhythmia is an established therapy. It is routinely used for patients with cardiac rhythm management devices and the risk of device and lead affectation is deemed to be low. This assumption is currently not supported by substantial and current scientific data, mostly relying on older reports. No large, prospective trials with a population of patients with modern cardiac rhythm management devices exists.

Aim of the study The aim is to systematically include and follow all patients with cardiac rhythm management devices presenting for external electrical cardioversion, to analyse the effects of external electrical cardioversion on leads and devices. Thereby, providing reliable evidence and detecting possible SAE with a low incidence. Furthermore, to gather information on efficacy and recurrence rate in this population, to examine the value of external electrical cardioversion for rhythm control in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed, written consent
* Atrial or ventricular arrhythmia with indication for CV
* Status post CRM implantation, including CRT-D

Exclusion Criteria:

* Age < 18 years
* Patients under guardianship or with mental disorders / disabilities
* lead implantation < 4 weeks prior to CV
* contraindications for eCV or transoesophageal echocardiographie (TOE)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with implanted cardiac rhythm devices (pacemakers, ICD and CRT)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite safety endpoint: Changes of lead and device parameters | 2 weeks after CV
  assessed by device interrogation, if any of the following criteria is met:
  * a rise in threshold (at constant pulse duration) of >1V
  * exit block of any of the pacing leads
  * loss of programming of the device
  * rise in shock impedance by 50%
  * rise in charge time by 50%
  * drop in battery voltage of ≥0.2V within < 6 weeks

SECONDARY OUTCOMES:
Efficacy Endpoint | within 15 minutes after CV
  Assessed by device interrogation and 12-lead ECG:
  - restoration of normal sinus rhythm after CV
Late changes of lead parameters | 2 weeks after CV
  Any of the below, assessed by device interrogation:
  * Lead impedance > 1000 Ohm
  * a rise in lead impedance by 50%
  * ventricular lead sensing < 2mV
  * atrial lead sensing < 1mV
Inadvertent induction of ventricular fibrillation | 10 seconds after CV
  Assessed by 3 lead monitoring ECG
Composite endpoint: Early lead changes | within 15 minutes after CV
  assessed by device interrogation, if any of the following criteria is met:
  * a rise in threshold (at constant pulse duration) of >1V
  * exit block of any of the pacing leads
  * Lead impedance > 1000 Ohm
  * a rise in lead impedance by 50%
  * ventricular lead sensing < 2mV
  * atrial lead sensing < 1mV
Loss of programming | within 15 minutes after CV
  assessed by device interrogation:
  - loss of programming of the device
Change of shock impedance | within 15 minutes after CV
  assessed by device interrogation:
  - rise in shock impedance by 50%
Change of charge time | within 15 minutes after CV
  assessed by device interrogation:
  - rise in charge time by 50%

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lüker, Dr., Principal Investigator — University Hospital Cologne; Daniel Steven, Prof. Dr., Study Director — University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, Germany